CLINICAL TRIAL: NCT02492295
Title: Low-dose Propofol for the Treatment of Severe Refractory Migraine Headache in the Emergency Department
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to logistic reason
Sponsor: Albert Einstein Healthcare Network (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HN4616
Record Dates: First submitted 2015-03-25; First posted 2015-07-08 (Estimated); Results first posted 2020-03-19 (Actual); Last update posted 2020-03-19 (Actual); Status verified 2017-05

CONDITIONS: Migraine Headache
MeSH Terms: conditions — Migraine Disorders | interventions — Propofol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Propofol (Experimental): Propofol is administered intravenously as a 0.5mg/kg (at a concentration of 10mg/mL, rounded to the nearest 0.5mL) initial bolus, followed by repeat 0.25mg/kg boluses (same rounding) every three to five minutes as needed to maintain RASS target -2 ("light sedation - awakens to voice <10 seconds") to RASS target of -3 ("moderate sedation - movement or eye opening without eye contact") for 15 minutes.
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Propofol — Propofol will be administered as a 0.5mg/kg (at a concentration of 10mg/mL, rounded to the nearest 0.5mL) initial bolus, followed by repeat 0.25mg/kg boluses (same rounding) every three to five minutes as needed to maintain RASS target -2 ("light sedation - awakens to voice <10 seconds") to RASS target of -3 ("moderate sedation - movement or eye opening without eye contact") for 15 minutes. No more than 1.5mg/kg of propofol will be administered over this time period. After the sedation session is complete, patients will be allowed to wake up and will be monitored in the ED for at least another hour prior to discharge.
  Other Names: Diprivan; Propoven

SUMMARY:
Migraine headache is a frequent Emergency Department complaint. While first-line Emergency Department treatment for this condition is well-established, optimal second-line treatment options are not well-defined. First line Emergency Department treatments include Non-Steroidal Anti-Inflammatory Drugs (NSAIDs), dopamine antagonists. Second line treatments that have been proposed include triptans, steroids, antiepileptics, benzodiazepines, magnesium and narcotics, but none have shown reliable Emergency Department efficacy (less than 50% in most studies). In the past ten years there have been several case series published on using low, sub-anesthetic doses of propofol for the treatment of refractory migraine. These case series have reported very impressive efficacy rates, especially in comparison to the published efficacy rates of other second-line treatments. Personal experience using this treatment modality has also yielded impressive clinical results. Most of the published series, however, have not been conducted in the Emergency Department.

The Investigators propose to conduct a prospective, observational trial of low-dose propofol for the treatment of refractory migraine in the Emergency Department. Propofol is a frequently-used Emergency Department sedative, with a good safety profile when administered by experienced Emergency Medicine practitioners using appropriate monitoring. The primary outcome measurement will be reduction of pain after treatment, with secondary outcome measures related to the safety of treatment and continuation of pain relief after leaving the Emergency Department. Although the protocol will involve the use of low-dose propofol with the aim of achieving light-to-moderate sedation only, all patients will care for and monitor at a level appropriate for deep procedural sedation.

DETAILED DESCRIPTION:
This is a prospective, open-label, observational trial to assess basic efficacy and safety in the Emergency Department treatment environment.

Emergency Department patients at Einstein Medical Center Philadelphia, with migraine type headache (International Headache Classification), who continue to have severe (6/10 or greater) pain one hour after receiving adequate first-line treatment with a dopamine antagonist (prochlorperazine or metoclopramide) and an NSAID (ketorolac or ibuprofen) will be approached for possible inclusion. Patients who meet all inclusion/exclusion criteria will be given informed consent, including consent for procedural sedation. Patients who decline to participate will continue to have their headache treated by the ED team as per usual practice.

After enrollment, patients will be set up for procedural sedation per standard Emergency Department protocol. This includes a well-running peripheral IV; continuous monitoring with telemetry, pulse oximetry, capnography and automated blood pressure checks; continuous bedside monitoring by both an Emergency Department nurse and an Emergency Department attending or senior resident (with immediate attending availability); and airway management tools including suction, oxygen, and Bag valve mask ventilation at bedside, with advanced airway management tools (intubation equipment, etc) immediately available. After time-out, propofol administration will begin. The study drug will be administered only by those properly trained to do so and will be administered in compliance with healthcare licensure requirements. Propofol will be administered as a 0.5mg/kg (at a concentration of 10mg/mL, rounded to the nearest 0.5mL) initial bolus, followed by repeat 0.25mg/kg boluses (same rounding) every three to five minutes as needed to maintain Richmond Agitation Sedation Scale (RASS) target -2 ("light sedation - awakens to voice <10 seconds") to RASS target of -3 ("moderate sedation - movement or eye opening without eye contact") for 15 minutes. No more than 1.5mg/kg of propofol will be administered over this time period. After the sedation session is complete, patients will be allowed to wake up and will be monitored in the ED for at least another hour prior to discharge.

If a patient experiences any adverse safety event that in the determination of the treating provider make it unsafe to continue giving propofol, the protocol will be terminated immediately.

Numeric pain score (0-10) will be obtained prior to medication administration, at 30 minutes and at 60 minutes after the final dose of medication. Patients will also be questioned about associated migraine symptoms (nausea/vomiting/photophobia/phonophobia) and their resolution. Patients will receive follow-up phone calls at 24 hours to assess pain score, need for additional medications and whether they would opt for the same treatment again in the event of another severe headache. Patient charts will subsequently be reviewed to determine if they had any further ED visits within 72 hours after propofol administration.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65
* Chief complaint consistent with the diagnosis of headache that meets 2 of the 4 following criteria (check all that apply):
* Unilateral Headache
* Pulsatile Sensation
* Moderate to Severe pain intensity
* Aggravation by physical activity or causing avoidance of physical activity (i.e. climbing stairs, walking)
* Headache is associated with at least one of the following symptoms (check all that apply):
* Nausea and/or vomiting
* Photophobia and/or phonophobia
* History of at least 5 similar headaches
* Within 6 hours of screening has received BOTH (via IV or PO):

  1. A Non-Steroidal Anti-Inflammatory Drug (NSAID):

     Ibuprofen / "Motrin" Naproxen / "Aleve" Ketorolac / "Toradol"
  2. A Dopamine-Antagonist:

Metoclopramide / "Reglan" Prochlorperazine / "Compazine"

* Persists with 6/10 or greater pain at one hour after above treatment
* Emergency Department attending feels patient appropriate for propofol treatment

Exclusion Criteria:

* Allergy to the study medication / eggs / soy (medication components)
* Inability to provide written, informed consent
* Employee or in police custody
* Pregnant or breast-feeding
* Medical concerns: Chronic obstructive pulmonary disease, active asthma exacerbation, obstructive sleep apnea, morbid obesity (Body Mass Index > 40), American Society of Anaesthesiologists class 3 or greater, actively intoxicated, Blood Pressure < 110/70
* Meal or heavy snack within 3 hours of sedation time
* Will be driving themselves home from Emergency Department
* Opioid use within the last 6 hours
* Previously enrolled in this study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2016-01-01 (Actual); Study Completion 2016-01-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Gardner, MD, Principal Investigator — Albert Einstein Health Network
Locations (1):
- Albert Einstein Medical Center, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 0 Participants analyzed. PI has left the institution. Efforts made to contact were unsuccessful. No data available
Pre-assignment Details: 0 Participants analyzed. PI has left the institution. Efforts made to contact were unsuccessful. No data available
Period: Overall Study
Arm/Group | Propofol
Started | 0
Completed | 0
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: 0 Participants analyzed. PI has left the institution. Efforts made to contact were unsuccessful. No data available
Groups:
- Propofol: Propofol: Propofol will be administered as a 0.5mg/kg (at a concentration of 10mg/mL, rounded to the nearest 0.5mL) initial bolus, followed by repeat 0.25mg/kg boluses (same rounding) every three to five minutes as needed to maintain RASS target -2 ("light sedation - awakens to voice <10 seconds") to RASS target of -3 ("moderate sedation - movement or eye opening without eye contact") for 15 minutes. No more than 1.5mg/kg of propofol will be administered over this time period. After the sedation session is complete, patients will be allowed to wake up and will be monitored in the ED fo
Arm/Group | Propofol
Number analyzed (Participants) | 0
Age, Categorical
Age, Continuous
Sex: Female, Male
Region of Enrollment [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: Pain Assessed by Numeric Pain Score
Description: Numeric pain score 1 hour after completion of propofol administration.
Time Frame: 60 minutes
Population: 0 Participants analyzed. PI has left the institution. Efforts made to contact were unsuccessful. No data available
Groups:
- Propofol: Propofol is administered intravenously as a 0.5mg/kg (at a concentration of 10mg/mL, rounded to the nearest 0.5mL) initial bolus, followed by repeat 0.25mg/kg boluses (same rounding) every three to five minutes as needed to maintain RASS target -2 ("light sedation - awakens to voice <10 seconds") to RASS target of -3 ("moderate sedation - movement or eye opening without eye contact") for 15 minutes.
  Pr
Arm/Group | Propofol
Number analyzed (Participants) | 0

2. Secondary Outcome: Pain Assessed by Numeric Pain Score
Description: Numeric Pain Score
Time Frame: 24 hours
Population: 0 Participants analyzed. PI has left the institution. Efforts made to contact were unsuccessful. No data available
Arm/Group | Propofol
Number analyzed (Participants) | 0

3. Secondary Outcome: Pain Assessed by Numeric Pain Score
Description: Numeric pain score 30 minutes after completion of propofol administration.
Time Frame: 30 minutes
Population: 0 Participants analyzed. PI has left the institution. Efforts made to contact were unsuccessful. No data available
Arm/Group | Propofol
Number analyzed (Participants) | 0

4. Secondary Outcome: Additional Rescue Medications Used
Description: Need for other pain relief medications for migraine after use of propofol
Time Frame: 24 hours
Population: 0 Participants analyzed. PI has left the institution. Efforts made to contact were unsuccessful. No data available
Arm/Group | Propofol
Number analyzed (Participants) | 0

5. Secondary Outcome: Patient Willingness to Use Propofol Again in Case of Refractory Migraine as Assessed by Patient Questionaire
Description: Assessed by questionnaire read to patient over phone (yes/no answer)
Time Frame: 24 hours
Population: 0 Participants analyzed. PI has left the institution. Efforts made to contact were unsuccessful. No data available
Arm/Group | Propofol
Number analyzed (Participants) | 0

6. Secondary Outcome: Emergency Room Re-admissions
Description: May reflect treatment failure or occurrence of adverse events/reactions-determined by Response is Yes or No
Time Frame: 72 hours
Population: 0 Participants analyzed. PI has left the institution. Efforts made to contact were unsuccessful. No data available
Arm/Group | Propofol
Number analyzed (Participants) | 0

7. Secondary Outcome: Hypoxia: SpO2 of <88%
Description: SpO2 of <88% up to 60 minutes after propofol administration or until patient is fully alert.
Time Frame: 60 minutes
Population: 0 Participants analyzed. PI has left the institution. Efforts made to contact were unsuccessful. No data available
Arm/Group | Propofol
Number analyzed (Participants) | 0

8. Secondary Outcome: Hypotension: Blood Pressure of < 100/60
Description: Blood pressure of < 100/60 up to 60 minutes after propofol administration or until patient is fully alert.
Time Frame: 60 minutes
Population: 0 Participants analyzed. PI has left the institution. Efforts made to contact were unsuccessful. No data available
Arm/Group | Propofol
Number analyzed (Participants) | 0

9. Secondary Outcome: Number of Patients Needing Basic Airway Repositioning Maneuver During Sedation
Description: Assessed by questionaire filled out by research associate during drug administration. This Will report the number of patients who required a basic airway repositioning maneuver (jaw thrust/head tilt) during the course of the sedation.
Time Frame: 60 minutes
Population: 0 Participants analyzed. PI has left the institution. Efforts made to contact were unsuccessful. No data available
Arm/Group | Propofol
Number analyzed (Participants) | 0

10. Secondary Outcome: Number of Patients Needing Advanced Airway Intervention (Beyond Simple Repositioning)(Composite)
Description: Assessed by questionnaire filled out by research associate during drug administration. Will report the composite number of patients (if any) who required an advanced airway maneuver, specifically insertion of a nasal-pharyngeal airway (NPA) or oro-pharyngeal airway (OPA), use of a bag-valve-mask (BVM), endotracheal intubation (ETT) or surgical airway. While only a composite number will be reported as a secondary outcome, we will give details in the text of any such interventions. We *do not* anticipate that any such interventions will be required during the study, and thus are not going to pre-specify the above interventions as separate individual outcome measures, but will instead report a composite number, with relevant details in the text.
Time Frame: 60 minutes
Population: 0 Participants analyzed. PI has left the institution. Efforts made to contact were unsuccessful. No data available
Arm/Group | Propofol
Number analyzed (Participants) | 0

11. Secondary Outcome: Number of Patients With Allergic (Anaphylactic-spectrum) Reactions That May be Attributed to Propofol Use (Composite)
Description: Assessed by questionnaire filled out by research associate during and after drug administration. The number of patients (if any) with an anaphylactic-spectrum response will be reported as a composite number, and in the text we will provide a specific description of the reaction(s), which might include itching, urticaria, airway swelling, or wheezing/stridor. Please note that we *do not* anticipate any such reactions to propofol, and thus are not going to pre-specificy these reactions individually as separate outcome measures, but will instead report a composite, with relevant details in the text.
Time Frame: 60 minutes
Population: 0 Participants analyzed. PI has left the institution. Efforts made to contact were unsuccessful. No data available
Arm/Group | Propofol
Number analyzed (Participants) | 0

12. Secondary Outcome: Hypercarbia: End Tidal Carbon Dioxide (ETCO2) of >50 mm Hg
Description: ETCO2 of >50 mm Hg up to 60 minutes after propofol administration or until patient is fully alert.
Time Frame: 60 minutes
Population: 0 Participants analyzed. PI has left the institution. Efforts made to contact were unsuccessful. No data available
Arm/Group | Propofol
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 0
Description: 0 Participants analyzed. PI has left the institution. Efforts made to contact were unsuccessful. No data available
Arm/Group | Propofol
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
0 Participants analyzed. PI has left the institution. Efforts made to contact were unsuccessful. No data available

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes